CLINICAL TRIAL: NCT01254357
Title: Burn Outcomes in Young Adult Burn Survivors- A Multicenter Outcomes Study
Brief Title: Burn Outcomes in Young Adult Burn Survivors
Acronym: YA
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Colleen Ryan, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2010P002459
Record Dates: First submitted 2010-11-29; First posted 2010-12-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Burns; Trauma
Keywords: Burns; Trauma; Outcomes; Quality of Life
MeSH Terms: conditions — Burns; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- YA Burned Subjects: Any person between the years of 19-30 years old treated for a burn injury, having incurred within past 12 months.
  Interventions: Other: Questionnaire self report

INTERVENTIONS:
Other: Questionnaire self report — Burn specific outcome measurement and global health measurement
  Other Names: Young Adult Burn Outcomes Questionnaire; Veterans Rand 12 Item Health Survey

SUMMARY:
As part of Clinical Trials.Gov ID:NCT00253292 a psychometrically sound outcomes instrument was developed to study the outcomes of burn survivors in the 19-30 year old age group. This workgroup has come together to re-examine the data collected during the previous study and determine next steps in understanding the recovery for this population.

DETAILED DESCRIPTION:
This study looks to understand previously collected outcomes scores. Identifying young adult burned patients at risk for poor outcomes remains an under-published field of study. We strive to identify problem areas for this population before they adversely effect their quality of life. How are these 19-30 year olds different from their non-burned counterparts and what interventions can we provide to equalize the balance?

ELIGIBILITY:
Inclusion Criteria:

All burn injured young adults with or without skin grafting. All burned young adults on or after their 18th birthday. Between the ages of 19-30 years. English speaking Present for inpatient or outpatient treatment. -

Exclusion Criteria:

Non-burn skin conditions. Non-English speaking young adults. Young adults less than 19 years of age. Young adults greater than 30 years of age.

-

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Persons having suffered a burn injury and treated at participating study sites that are between the ages of 19-30 years of age and speak English.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Short Form Young Adult Outcomes Questionnaire | 12-24 month follow-up
  Once existing data are massaged we will revise the stated outcome measure to make it more contemporary.

SECONDARY OUTCOMES:
Veterans Rand 12 Item Health Survey (VR-12) | 12-24 months follow-up
  The VR-12 instrument was developed based on data from the SF-36 survey.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Ryan, MD, Principal Investigator — Shriners Hospitals for Children and Massachusetts General Hospital; Jeffrey Schneider, MD, Study Director — Massachusetts General Hospital and Spaulding Rehab Hospital; Tina Palmieri, MD, Study Director — Shriners Hospitals or Children,University of CA at Davis; David Herndon, MD, Study Director — Shriners Hospitals forChildren, University of TX Medical Branch; Lewis Kazis, ScD, Study Chair — Shriners Hospitalsfor Children, Boston University School of Public Health; Ronald G Tompkins, MD, Study Director — Shriners Hospitals for Children, Massachusetts General Hospital
Locations (6):
- United States (6):
  - Shriners Hospital for Children, Sacramento, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Mass General Hospital, Boston, Massachusetts
  - Shriners Hospital for Children - Boston, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Shriners Hospital for Children - Galveston, Galveston, Texas